CLINICAL TRIAL: NCT06045715
Title: An Optimized Post-surgery Follow-up Strategy for Patients With Esophageal Cancer
Brief Title: Follow-up Strategy for Esophageal Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jianhua Fu, Professor, Sun Yat-sen University
Other Study IDs: 20220820
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-09

CONDITIONS: Esophagus Cancer
Keywords: follow-up
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- follow-up: patients were follow-up with different time intervals
  Interventions: Other: follow-up with different time intervals

INTERVENTIONS:
Other: follow-up with different time intervals — After radical surgery, patients are followed up with different time intervals

SUMMARY:
The recurrence risk of patients with esophageal cancer was stratified by integrating different stages and pathological factors. The risk of recurrence was dynamically estimated for each group of patients, and the optimal follow-up strategy was developed based on the recurrence risk.

DETAILED DESCRIPTION:
Patients with histologically proven, esophageal cancer (EC) patients diagnosed between 2008 and 2018 were recruited. Recursive partition analysis was applied to develop recurrence risk stratification for patients. The follow-up strategies of each stratification were developed based on monthly recurrence probability and validated by bootstrap validation and an external dataset. Markov decision-analytic models were constructed to evaluate the cost-effectiveness of the follow-up strategies.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients aged between 18 and 80 years old; (2) Pathological diagnosis as esophageal squamous cell carcinoma or adenocarcinoma; (3) Patients underwent esophagectomy and received R0 resection.

Exclusion Criteria:

(1) Patients with secondary primary tumor; (2) Patients who died within 30 days after surgery or died of post-operation complications; (3) Patients missing essential clinical information, such as operation record, pathological diagnosis, and follow-up data; (4) Patients with radiologically or histologically confirmed distant metastasis; (5) Patients previously underwent endoscopic mucosal resection or definitive radiochemotherapy as initial treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with historically proven esophageal squamous cell carcinoma and adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 2008-2020
  disease-free survival

SECONDARY OUTCOMES:
local relapse-free survival | 2008-2020
distant metastasis-free survival | 2008-2020

CONTACTS AND LOCATIONS:
Locations (1):
- Jianhua Fu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Due to the policy, we could not shared the data